CLINICAL TRIAL: NCT01386853
Title: A 12-week, Randomized, Multicenter, Double-blind, Active-controlled, Non-inferiority Study to Compare the Efficacy and Safety of Pitavastatin and Atorvastatin in High Risk Hypercholesterolemic Patients
Brief Title: Efficacy and Safety Study of Pitavastatin and Atorvastatin in High Risk Hypercholesterolemic Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tai Tien Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Manager, Development Department
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TATPITA20101005
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; Pitavastatin; Atorvastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin (Experimental)
  Interventions: Drug: Pitavastatin
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — 2 mg QD
  Other Names: Livalo
  Arms: Pitavastatin
Drug: Atorvastatin — 10 mg QD
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
This is a 12-week, randomized, multicenter, double-blind, active-controlled, non-inferiority study (TATPITA20101005) to compare the efficacy and safety of pitavastatin (Livalo®) and atorvastatin (Lipitor®) in high risk hypercholesterolemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 20 years old and < 75 years old.
* Patient who was eligible and able to participate in the study and accepts to enter the study by signing written informed consent.
* Patient with fasting LDL-C > 100 mg/dL. The concentration of LDL-C is obtained from laboratory examination.
* Patient with at least one of the following description (NCEP ATP III guideline).
* Female patient with child-bearing potential must take reliable contraception method(s) during the participation of the study.

Exclusion Criteria:

* Patient who has participated in other investigational studies within 3 months.
* Patient took medication and natural health foods known to alter blood lipid profiles within 4 weeks.
* Patient is taking any medication or food that is prohibited by the study.
* Patient taking Amiodarone will be excluded from this study (due to long half life of this medication).
* Patient is diagnosed with type 1 DM or has been using insulin/insulin analog medication.
* Patient with a history of multiple drug allergies or with a known allergy to HMG-CoA reductase inhibitors.
* Patient with TG > 400 mg/dL.
* Excessive obesity defined as BMI above 35 kg/m2.
* Cerebral vascular disease (including cerebrovascular hemorrhage or ischemia, transient ischemic attack) diagnosed within 3 months.
* Myocardial infarction, heart failure (NYHA class III or IV), gross cardiac enlargement (cardiothoracic ratio > 0.5), significant heart block or cardiac arrhythmias within 3 months; history of uncontrolled complex ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardia, pacemaker or implantable cardiac device were not eligible for this study.
* Patient with advanced renal disorder (Serum creatinine levels ≥ 2 mg/dL and BUN ≥ 25 mg/dL).
* Patient with advanced hepatic disorder (AST or ALT level ≥ 100 IU/L)
* Patient with CK level > 5 × ULRR at any time point between Visit 1 and Visit 2.
* Patient with poorly controlled diabetes mellitus (HbA1c > 9.0%) or patient with severe hypertension (> 180 mmHg for systolic or > 120 mmHg in diastolic blood pressure).
* Patient with hypothyroidism, hereditary muscular disorders, family history of the above or history of drug-induced myopathy.
* Patient has significant alcohol consumption (> 65 mL pure alcohol) within 48 hours before Visit 2.
* Any major surgery within 3 months prior to Visit 2.
* Female patient who is lactating, being pregnant or plans to become pregnant.
* Patient with conditions judged by the investigator as unsuitable for the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The change of LDL-C | Baseline to 12 weeks

SECONDARY OUTCOMES:
The proportion of patients achieving LDL-C < 100 mg/dL; the changes of HDL-C, TG, non-HDL-C, Apo A1 and Apo B, fasting plasma glucose, fasting insulin level, insulin resistance by the HOMA-IR, HbA1c, free fatty acid, and ADMA | Baseline to 4 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Wen Chen, M.D. Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taipei, Taiwan
Locations (6):
- Taiwan (6):
  - Changhua Christian Hospital, Chang-hua
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Memorial Hospital-LinKou, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Derived] Lin LY, Huang CC, Chen JS, Wu TC, Leu HB, Huang PH, Chang TT, Lin SJ, Chen JW. Effects of pitavastatin versus atorvastatin on the peripheral endothelial progenitor cells and vascular endothelial growth factor in high-risk patients: a pilot prospective, double-blind, randomized study. Cardiovasc Diabetol. 2014 Jul 16;13:111. doi: 10.1186/s12933-014-0111-1. PMID 25027585
- [Derived] Liu PY, Lin LY, Lin HJ, Hsia CH, Hung YR, Yeh HI, Wu TC, Chen JY, Chien KL, Chen JW. Pitavastatin and Atorvastatin double-blind randomized comPArative study among hiGh-risk patients, including thOse with Type 2 diabetes mellitus, in Taiwan (PAPAGO-T Study). PLoS One. 2013 Oct 1;8(10):e76298. doi: 10.1371/journal.pone.0076298. eCollection 2013. PMID 24098467